CLINICAL TRIAL: NCT03369080
Title: Prospective Representative National Survey of Body Mass Index in People With Spinal Cord Injury.
Brief Title: Prospective Survey of Body Mass Index in People With Spinal Cord Injury.
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Metropolitan University College (Other); Spinal Cord Injury Centre of Western Denmark (Other)
Responsible Party: Principal Investigator, Nicolaj Jersild Holm, Ph.D student, Rigshospitalet, Denmark
Other Study IDs: sub project 1
Record Dates: First submitted 2017-11-17; First posted 2017-12-11 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
Keywords: Body Mass Index
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish National Cohort: This study includes all patients with a new Spinal Cord Injury hospitalized at Clinic for Spinal Cord Injuries, Rigshospitalet or Spinal Cord Injury Center of Western Denmark

SUMMARY:
This study is a prospective national survey of body mass index, and includes all patients with a new spinal cord injury hospitalized at Clinic for Spinal Cord Injuries, Rigshospitalet and Spinal Cord Injury Center of Western Denmark during a period of 9 months. Informed consent is retrieved from all participants.

DETAILED DESCRIPTION:
The current study is a sub- study in a Ph.D project containing 4 sub- studies. The protocol for the current study includes all four sub- studies, and each of the other three sub- studies will be registered ongoing individually. The current study is a prospective national survey of body mass index (BMI), and includes all patients with a new spinal cord injury hospitalized at Clinic for Spinal Cord Injuries, Rigshospitalet (CSCI) and Spinal Cord Injury Center of Western Denmark during a period of 9 months whereby 100 patients are expected to participate. Data are collected at admission and discharge. At CSCI BMI is collected every 6 weeks and all outcome measures will also be collected at follow up 6 months after discharge. A VO2peak test at discharge is performed as well, and in some participants accelerometry is performed in order to describe the amount and intensity of physical activity. Test- retest reliability of the VO2peak test and accelerometry is investigated as well. Patients with a new Spinal Cord Injury within the last 12 months, who are admitted for rehabilitation several months after the time of injury are also included in the prospective survey. Therefore the data for BMI at the time of injury is collected for all patients at admission to primary rehabilitation from both the patient journal and also by asking the patient about weight and height at the time of injury

ELIGIBILITY:
Inclusion Criteria:

* All newly injured patients with Spinal Cord Injury (within the last 12 months)admitted at Clinic for Spinal Cord Injuries, Rigshospitalet and Spinal Cord Injury Centre of Western Denmark, are included regardless of age, neurological level of lesion and completeness of the injury if informed consent is retrieved.

Exclusion Criteria:

* Insufficient skills in Danish language
* Reduced mental function that prevents reading and answering the questionnaires

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All newly injured patients with Spinal Cord Injury admitted at Clinic for Spinal Cord Injuries, Rigshospitalet and Spinal Cord Injury Centre of Western Denmark
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Change from baseline to follow-up 6 months after discharge from primary rehabilitation
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2

OTHER OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury | At admission
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. The International Standards for Neurological Classification of Spinal Cord Injury defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded according to the American Spinal Injury Association Impairment Scale
International Standards for Neurological Classification of Spinal Cord Injury | At discharge in average 4-6 months after admission to primary rehabilitation
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. TheInternational Standards for Neurological Classification of Spinal Cord Injury defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded according to the American Spinal Injury Association Impairment Scale
International Standards for Neurological Classification of Spinal Cord Injury | At follow up 6 months after discharge
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. The International Standards for Neurological Classification of Spinal Cord Injury defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded according to the American Spinal Injury Associationment Impairment Scale
Spinal Cord Injury Independence Measure III | At admission
  The Spinal Cord Injury Independence Measure III is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Spinal Cord Injury Independence Measure III | At discharge in average 4-6 months after admission to primary rehabilitation
  The Spinal Cord Injury Independence Measure III is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Spinal Cord Injury Independence Measure III | At follow up 6 months after discharge
  The Spinal Cord Injury Independence Measure III is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Patient Health Questionnaire- 2 | At admission
  The Patient Health Questionnaire- 2 comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
Patient Health Questionnaire- 2 | At discharge in average 4- 6 months after admission to primary rehabilitation
  Patient Health Questionnaire- 2 comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
Patient Health Questionnaire- 2 | At follow up 6 months after discharge
  The Patient Health Questionnaire- 2 comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
The International SCI Quality of Life Basic Data Set | At admission
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological health
The International SCI Quality of Life Basic Data Set | At discharge in average 4- 6 months after admission to primary rehabilitation
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological health
The International SCI Quality of Life Basic Data Set | At follow up 6 months after discharge
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological health
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury ( | At admission
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury ( | At discharge in average 4-6 months after admission to primary rehabilitation
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury ( | At follow up 6 months after discharge
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At admission
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At discharge in average 4-6 months after admission to primary rehabilitation
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At follow up 6 months after discharge
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
VO2peak | At discharge in average 4- 6 months after admission to primary rehabilitation
  Measures the maximal oxygen consumption in ml/kg/min
Objective physical activity (accelerometry) | At discharge in average 4- 6 months after admission to primary rehabilitation
  Is measured with a multisensor device recording accelerations and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaj J Holm, Ph.D student, Principal Investigator — Rigshopitalet, Clinic for Spinal Cord Injuries
Locations (1):
- Clinic for Spinal Cord Injuries, Rigshopitalet, Hornbæk, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holm NJ, Moller T, Adamsen L, Dalsgaard LT, Biering-Sorensen F, Schou LH. Health promotion and cardiovascular risk reduction in people with spinal cord injury: physical activity, healthy diet and maintenance after discharge- protocol for a prospective national cohort study and a preintervention- postintervention study. BMJ Open. 2019 Dec 31;9(12):e030310. doi: 10.1136/bmjopen-2019-030310. PMID 31892644

DOCUMENTS (1):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT03369080/Prot_000.pdf